CLINICAL TRIAL: NCT02306629
Title: An Open-label, Parallel-group, Single-dose Escalation Study to Evaluate the Pharmacokinetics, Safety, Tolerability and Pharmacodynamics of Subcutaneous Epratuzumab in Healthy Caucasian and Japanese Subjects
Brief Title: Study to Compare Properties of Epratuzumab When Given as an Injection Under the Skin or Directly Into the Blood
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Biopharma S.P.R.L. (Industry)
Collaborators: Pharmaceutical Research Associates (Other); Richmond Pharmacology Limited (Industry); ACM Global Laboratories (Other); Eurofins (Industry); The Doctors Laboratory Ltd (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SL0032; 2014-000911-15 (EudraCT Number)
Record Dates: First submitted 2014-11-29; First posted 2014-12-03 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Epratuzumab dose 1 sc (Experimental): This group of Caucasian and Japanese subjects will receive one single dose 1 of epratuzumab subcutaneous
  Interventions: Biological: Epratuzumab sc
- Epratuzumab dose 2 sc (Experimental): This group of Caucasian and Japanese subjects will receive one single dose 2 of epratuzumab subcutaneous
  Interventions: Biological: Epratuzumab sc
- Epratuzumab dose 3 sc (Experimental): This group of Caucasian subjects will receive one single dose 3 of epratuzumab subcutaneous
  Interventions: Biological: Epratuzumab sc
- Epratuzumab dose 2 iv (Active Comparator): This group of Caucasian and Japanese subjects will receive one single dose 2 of epratuzumab as an intra venous infusion
  Interventions: Biological: Epratuzumab iv

INTERVENTIONS:
Biological: Epratuzumab sc — Active substance: Epratuzumab, Pharmaceutical form: Solution for injection, Route of Administration: Subcutaneous,
  Arms: Epratuzumab dose 1 sc; Epratuzumab dose 2 sc; Epratuzumab dose 3 sc
Biological: Epratuzumab iv — Active substance: Epratuzumab, Pharmaceutical form: Solution for Infusion, Route of Administration: Intravenous,
  Other Names: CDP3194; EMAB
  Arms: Epratuzumab dose 2 iv

SUMMARY:
To assess how the absolute bioavailability, dose proportionality, pharmacokinetics, safety and tolerability of epratuzumab compared when given as a subcutaneous (sc) injection as to when given as an intravenous (iv) infusion in Caucasian and Japanese healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female.
* At the Screening Visit, subject is 18 years to 50 years, inclusive (for Caucasian subjects), or 20 years to 50 years (for Japanese subjects)
* Subject must be in good health (physically and mentally) as determined by the investigator on the basis of medical history
* Subject has a body weight of 45 kg to 90 kg, inclusive, and body mass index (BMI) between 18.0 kg/m2 and 29.9 kg/m2, inclusive
* Japanese subjects are defined as a person carrying a Japanese passport, who is a descendant of 4 Japanese grandparents and has not been outside Japan for more than 5 years prior to screening
* Females of childbearing potential are required to have a negative serum pregnancy test at the Screening Visit and must agree to use an acceptable method of birth control during the study and for a period of 3 months after the administration of investigational medicinal product (IMP)
* Male subjects must agree to use an acceptable method of contraception during the study and for at least 3 months after receiving IMP unless they have undergone vasectomy

Exclusion Criteria:

* Subject has donated blood (including through participation in another clinical study) or suffered blood loss (≥450 mL) <60 days prior to dosing, or has donated platelets <14 days prior to dosing
* Subject has active malignancies or a history of malignancy
* Subject has a history of severe or multiple allergies
* Subject has a history of chronic infection, recent serious or life-threatening infection
* Subject with a recurrent history or active systemic/respiratory infection due to fungal, parasitic, or mycotic pathogens
* Subject has a positive HBsAg, anti-HCV or anti-HIV test result during the Screening Period
* Subject has a history of or a concurrent clinically significant illness, medical condition, or laboratory abnormality that, in the investigator's opinion, could affect the safety of the subject upon exposure to epratuzumab or confound the results of the study
* Female subjects who are breast feeding, pregnant, or plan to become pregnant during the study or within 3 months following dosing of the IMP
* Subjects who are immunocompromised
* A confirmed positive urine drug screen
* Subject has a history of substance abuse, drug addiction, or alcoholism within 3 years prior to study admission
* Subject is unable or unwilling to stop smoking during the inpatient stay
* Subject has previous exposure to, or has participated in studies with, any other anti-B-cell therapies
* Subject has a medical condition that requires chronic medication
* Subject has received a live vaccine in the month prior to the administration of IMP or is scheduled or expected to receive live vaccines during the study period or for 3 months after administration of the IMP

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2014-11; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration time curve from Baseline to time of last detectable concentration (AUC(0-t)) | From Baseline (Day 1 pre-dose) to Day 85 (End of study)
Area under the plasma concentration time curve from zero up to infinity (AUC(0-inf)) | From Baseline (Day 1 pre-dose) to Day 85 (End of study)
Maximum observed plasma concentration (Cmax) | From Baseline (Day 1 pre-dose) to Day 85 (End of study)
Absolute bioavailability of the tested single sc doses | From Baseline (Day 1 pre-dose) to Day 85 (End of study)

SECONDARY OUTCOMES:
Time of observed Cmax (tmax) | From Baseline (Day 1 pre-dose) to Day 85 (End of study)
Apparent terminal half-life (t½) | From Baseline (Day 1 pre-dose) to Day 85 (End of study)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (1):
- 01, London, United Kingdom